CLINICAL TRIAL: NCT02975414
Title: Prospective Observational Cohort Study of Robot-assisted Laparoscopic Hernia Umbilical Hernia Repair (rTARUP)
Brief Title: Robotic Utility for Surgical Treatment of Umbilical Hernias
Acronym: Robust_2
Status: Completed | Type: Observational
Sponsor: Filip Muysoms (Other)
Responsible Party: Sponsor-Investigator, Filip Muysoms, surgeon, Algemeen Ziekenhuis Maria Middelares
Organization: Algemeen Ziekenhuis Maria Middelares (Other)
Other Study IDs: Robust_2
Record Dates: First submitted 2016-10-24; First posted 2016-11-29 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Hernia, Umbilical
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: rTARUP technique — obot-assisted rTARUP technique

SUMMARY:
The purpose of this study is the measurement of the evolution of the operation time during the start-up phase of robotic assisted surgery for the treatment of incisional hernia's of 40 patients treated in Maria Middelares in laparoscopic rTARUP technique.

DETAILED DESCRIPTION:
Minimally invasive hernia repair by laparoscopy is the standard treatment in adult patients with an umbilical hernia larger than 2 cm in Maria Middelares, Ghent.

As previously described in a chapter in a surgical guide and in a review article on the surgical fixation technique for laparoscopic umbilical hernia repair, the used technique has been proven feasible end safe.

Robot-assisted laparoscopic surgery has become standard in urology for resection of the prostate carcinoma. In general abdominal surgery, a large group of surgeons are currently working on the introduction of robotic-assisted surgery for resection of colon and rectal cancer in their daily practice. The third generation robot (DaVinci Xi), has extended the applicability of this technology within the field of general surgery.

For the surgical treatment of hernia's and other abdominal wall defects (umbilical or/and incisional hernia's), currently only surgeons in the US have experiences in structured treatment programs.

From September 1, 2016 Maria Middelares hospital will introduce robot-assisted surgery, including the laparoscopic TARUP umbilical hernia repair.

Main obstacles to the introduction of robot technology in abdominal wall surgery are prolonged preparation time in the operating room required for installation of the robot, and higher material costs related to the robot-assisted surgery. However, there are few precise data available on the exact size of extra time or increased costs related to the introduction of robotic assisted surgery in a program for abdominal surgery.

The purpose of this study is the measurement of the evolution of the operation time during the start-up phase of robotic-assisted surgery for the treatment of umbilical hernias by 40 patients in Maria Middelares hospital.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients selected and operated by the PI.

Exclusion Criteria:

* patients under the age of 18
* pregnancy
* no Informed Consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who are scheduled for laparoscopic repair of an umbillical hernia. A total of 40 patients will be enrolled in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
duration of operation | from the start of the operation until the end of the operation, approximately 4 hours
  Recording of the operation time needed for robot-assisted TARUP umbilical hernia repair

SECONDARY OUTCOMES:
intra-operative complications | until 4 weeks post-operative
  Intra-operative complications registered until 4 weeks after the hernia repair
post-operative complications | until 1 year post-operative
  Post-operative complications detected until 1 year after hernia repair by clinical follow up.
Questionnaire about the Quality of Life | until 1 year post-operative
  Quality of Life measured with the EuraHS QoL score preoperative and until 1 year after hernia repair by clinical follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, PhD, Principal Investigator — Maria Middelares hospital
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muysoms F, Van Cleven S, Pletinckx P, Ballecer C, Ramaswamy A. Robotic transabdominal retromuscular umbilical prosthetic hernia repair (TARUP): observational study on the operative time during the learning curve. Hernia. 2018 Dec;22(6):1101-1111. doi: 10.1007/s10029-018-1825-x. Epub 2018 Sep 22. PMID 30244344